CLINICAL TRIAL: NCT06443645
Title: Role of Sodium-glucose Linked Transporter 2 (SGLT2) and Its Inhibitor Over CARdiotoxicity Induced by Anthracyclines and Breast Cancer Tumorigenesis - SCARA-B
Brief Title: Role of Sodium-glucose Linked Transporter 2 (SGLT2) and Its Inhibitor Over CARdiotoxicity Induced by Anthracyclines and Breast Cancer Tumorigenesis SCARA-B
Acronym: SCARA-B
Status: Recruiting | Type: Observational
Sponsor: Centre Paul Strauss (Other)
Collaborators: Centre de Recherche en biomédecine de Strasbourg INSERM UMR-S1118 (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2023-024
Record Dates: First submitted 2024-05-13; First posted 2024-06-05 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Breast Neoplasms
Keywords: Breast cancer; Cardiotoxicities; SGLT2; Anthracyclines
MeSH Terms: conditions — Breast Neoplasms; Cardiotoxicity | interventions — Anthracyclines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adjuvant scheme: Indication for anthracycline-based chemotherapy after first-line surgery
  Interventions: Drug: Anthracycline
- Neoadjuvant scheme: Indication for anthracycline-based chemotherapy
  Interventions: Drug: Anthracycline

INTERVENTIONS:
Drug: Anthracycline — as standard of care

SUMMARY:
In the context of breast cancer, in case of an indication for chemotherapy, anthracycline-based protocols make it possible to improve the overall survival of patients most at risk. The frequency of anthracycline-related cardiac toxicities (ARCT) increases with the cumulative dose of anthracyclines administered and explains, at least in part, the increased risk of cardiovascular (CV) mortality in patient populations treated for breast cancer. The numerous indications for anthracycline-based protocols have made it possible to describe ARCT, among which heart failure with reduced left ventricular ejection fraction (LVEF) remains one of the most comorbid. In addition to left ventricular dysfunction, anthracyclines have been associated with endothelial dysfunction, microvascular damage and myocardial ischemia responsible for dilated cardiomyopathy.

Different approaches have attempted to better understand and prevent these ARCT. However, apart from the notion of limit cumulative doses of anthracyclines, few of them have made it possible to screen patients at risk and prevent the onset of cardiac dysfunction. The search for biological markers (Troponin I, BNP) or ultrasound markers (Longitudinal Strain) warning of subclinical cardiac damage is still struggling to assert its interest due in particular to significant inter- and intra-observer variability. Therapeutically, ACE inhibitors and beta-blockers have shown a significant improvement in the incidence rate of LVEF reduction during adjuvant treatment of breast cancer. However, despite equivalent signals in other cancers, the studies conducted to date are insufficiently powered and the role of these treatments is limited to secondary prevention or the treatment of objective heart failure. It remains necessary to determine new biological markers that can identify patients most at risk of ARCT and thus adapt our therapeutic prevention strategies. To do this, it is first necessary to better understand the pathophysiology underlying these ARCT.

The objective of this study is to determine whether expression of the receptor among endothelium and circulating cells, SGLT2, is associated with an additional risk of presenting cardiovascular toxicity following treatment with anthracycline. If this association is demonstrated, it will then be possible to better screen and prevent these cardiovascular complications.

ELIGIBILITY:
Inclusion Criteria:

* Patient > 18 years old
* Diagnosed with localized breast cancer
* Indication for first-line surgery or anthracycline-based chemotherapy.

Exclusion Criteria:

* History of chemotherapy or targeted therapy or immunotherapy administered before inclusion
* Patient currently being treated with anti-SGLT2, conversion enzyme inhibitor or ARA2
* Patient with known heart disease (ischemic, rhythmic, valvular, etc.)
* Patient with a Glomerular filtration rate < 45 mL/min/1.73m² according to the pre-therapeutic assessment
* Patient with impaired liver function
* Patient who is pregnant or breastfeeding
* Patient with a second cancer undergoing treatment
* Patient under guardianship or curatorship, protection of justice or deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The recruited population concerns adult patients followed for localized breast cancer and for whom treatment with anthracycline is indicated in the adjuvant or neoadjuvant situation.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-02-17 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate the expression of SGLT2 | At cycles 1, 2, 3, 4 and 2-3 weeks after end of treatement.
  Measurement of protein expression (Western Blot) and mRNA (RT-qPCR) of SGLT2 within the different models studied and according to the cumulative quantity of anthracyclines received and the patient's cardiovascular history before and after epirubine infusion.
Evaluate the expression of SGLT2 | At cycles 1, 2, 3, 4 and 2-3 weeks after end of treatement.
  Measurement of the polarization of peripheral blood mononuclear cells (PBMCs) into pro-inflammatory M1 and anti-inflammatory M2 before and after epirubine infusion.
Evaluate the expression of SGLT2 | At cycles 1, 2, 3, 4 and 2-3 weeks after end of treatement.
  Fluorescence measurement of the level of reactive oxygen species (ROS) formation and senescence of cardiovascular cells before and after epirubine infusion.
Evaluate the expression of SGLT2 | At cycles 1, 2, 3, 4 and 2-3 weeks after end of treatement.
  Measurement of inflammatory mediators secreted by circulating cells.Comparison with positive and negative controls that induce inflammation and ROS before and after epirubine infusion.

SECONDARY OUTCOMES:
Evaluate the ex vivo functional impact at the endothelial and cardiac level of exposure to patient plasma during treatment | At cycles 1, 2, 3, 4 and 2-3 weeks after end of treatement.
  Measurement of the antiplatelet activity of endothelial celles (ECs) mediated by nitric oxide (NO), the procoagulant activity and the adhesion of platelets and monocytes to ECs before and after epirubine infusion.
Evaluate the ex vivo functional impact at the endothelial and cardiac level of exposure to patient plasma during treatment | At cycles 1, 2, 3, 4 and 2-3 weeks after end of treatement.
  Quantification of inflammatory mediators in plasma and produced by treated cardiovascular cells before and after epirubine infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Hervé BISCHOFF, Principal Investigator — Centre Paul Strauss
Locations (1):
- Centre Paul Strauss, Strasbourg, France